CLINICAL TRIAL: NCT01090128
Title: Phase I Study of Neoadjuvant Chemotherapy With Nanoparticle Albumin Bound Paclitaxel, Doxorubicin and Cyclophosphamide (NAC) in Patients With Stages II-III Breast Cancer
Brief Title: Study of Neoadjuvant Chemotherapy With Nanoparticle Albumin Bound Paclitaxel, Doxorubicin and Cyclophosphamide (NAC) in Patients With Stages II-III Breast Cancer
Acronym: NAC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug Manufacturer withdrew support for studies not in metastatic breast cancer
Sponsor: University of Utah (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI53989
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Stages II-III Breast Cancer
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Nanoparticle Albumin Bound Paclitaxel; Drug: doxorubicin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: Nanoparticle Albumin Bound Paclitaxel — IV administered over 30 minutes. 100 mg/m2 on days 1 and 8
  Other Names: Abraxane
Drug: doxorubicin — 50 mg/m2 every 3 weeks
  Other Names: Adriamycin
Drug: cyclophosphamide — 500 mg/m2 given every 3 weeks

SUMMARY:
The purpose of this clinical trial is to test whether treatment of patients with breast cancer with the combination of Abraxane (nab-paclitaxel), Adriamycin (doxorubicin), and Cyclophosphamide prior to surgery is safe and results in good tumor response. Up to 24 patients may be enrolled in this study at the Mitchell Cancer Institute. All patients enrolling in this study will receive treatment with the combination of Abraxane, Adriamycin, and Cyclophosphamide.

DETAILED DESCRIPTION:
This is a single center, open phase I dose escalation study with expansion cohort. The dose escalation part of the study is now closed and the highest tolerable dose of nab-paclitaxel (Abraxane) was assessed to be 100 mg/m2 in combination with doxorubicin (Adriamycin) and cyclophosphamide in patients with stages II-III breast cancer in the neoadjuvant setting. The initial phase I study objective was to primarily assess the safety of the drug combination, and to secondarily obtain preliminary data on the clinical efficacy of the combination. 25 patients were enrolled. The expansion cohort will enroll 15 additional patients.

The purpose of the expansion cohort is to assess pathological complete response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven adenocarcinoma of the breast stages II-III, according to the AJCC Staging Manual, 7th Edition, 2009
2. The following receptor status:

   Expansion: Triple negative (ER<1%, PR<1%, and Her-2/neu negative Phase 1 (closed): Negative Her-2/neu status
3. ECOG performance status 0 or 1
4. Negative pregnancy test
5. Normal cardiac function (ejection fraction > lower limit of normal) as determined by MUGA or echocardiogram
6. ANC greater than or equal to 1,500/mm3; platelet greater than or equal to 100,000/mm3; hemoglobin greater than or equal to 9 gm/dL
7. Serum bilirubin levels less than or equal to 1.5 mg/dL
8. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) less than or equal to 2.5 X upper limit of normal, alkaline phosphatase less than or equal to 2.5 X upper limit of normal.
9. Serum creatinine levels less than or equal to 1.5 mg/dL
10. Women of childbearing potential should be advised to avoid becoming pregnant while receiving treatment with nab-paclitaxel through 28 days after the last dose. Men should be advised to not father a child while receiving treatment with azacitidine or nab-paclitaxel. Appropriate methods of birth controls for women include oral or implanted contraceptives, intrauterine device (IUD), diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner and also based on the judgment of the investigator.
11. Female, greater than or equal to 19 years of age and any race.

Exclusion Criteria:

1. Concurrent therapy with any other non-protocol anti-cancer therapy
2. For Phase I patients only: Current therapy with hormone replacement therapy, or any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators
3. Presence of neuropathy > grade 2 (NCI-CTC version 3.0) at baseline
4. History of any other malignancy requiring active treatment
5. Clinically significant cardiovascular disease (e.g., hypertension [BP > 150/100], myocardial infarction or stroke within 6 months, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
6. Currently active infection.
7. History of HIV infection or chronic hepatitis B or C.
8. The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications
9. Pregnancy or breast feeding
10. A history of a severe hypersensitivity reaction to nab-paclitaxel.
11. Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity, timing, seriousness and relatedness of adverse events and laboratory abnormalities | one year
Pathologic complete response | 1 year

SECONDARY OUTCOMES:
Overall clinical response rate (OcRR) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hung Khong, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Huntsman Cancer Institute, Salt Lake City, Utah, United States